CLINICAL TRIAL: NCT02790034
Title: A Randomised, Double-Blind, Placebo-Controlled 6-month Study to Evaluate the Efficacy, Safety, and Tolerability of Sarizotan in Patients With Rett Syndrome With Respiratory Symptoms
Brief Title: Evaluation of the Efficacy, Safety, and Tolerability of Sarizotan in Rett Syndrome With Respiratory Symptoms
Acronym: STARS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study did not demonstrate evidence of efficacy on the primary or secondary efficacy variables
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sarizotan/001/II/2015
Record Dates: First submitted 2016-05-24; First posted 2016-06-03 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — sarizotan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sarizotan low dose (Experimental): 2 mg or 5 mg bid based on age and weight criteria for 24 wks DB 2 mg bid (4 to <13 years; ≥13 years of age and weighing <25 kg 5 mg bid (≥13 years of age and weighing ≥25 kg)
  Interventions: Drug: Sarizotan low dose
- Sarizotan high dose (Experimental): 5 mg or 10 mg bid based on age and weight criteria for 24 wks DB 5 mg bid (4 to <13 years; ≥13 years of age and weighing <25 kg 10 mg bid (≥13 years of age and weighing ≥25 kg)
  Interventions: Drug: Sarizotan high dose
- Placebo (Placebo Comparator): Placebo bid for 24 wks DB age 4 and above
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sarizotan low dose — 2 mg or 5 mg bid based on age and weight criteria for 24 wks DB 2 mg bid (4 to <13 years; ≥13 years of age and weighing <25 kg; 5 mg bid (≥13 years of age and weighing ≥25 kg). Assessment of safety, tolerability and efficacy on reducing the respiratory symptoms in patients.
  Arms: Sarizotan low dose
Drug: Sarizotan high dose — 5 mg or 10 mg bid based on age and weight criteria for 24 wks DB 5 mg bid (4 to <13 years; ≥13 years of age and weighing <25 kg; 10 mg bid (≥13 years of age and weighing ≥25 kg) Assessment of safety, tolerability and efficacy on reducing the respiratory symptoms in patients
  Arms: Sarizotan high dose
Drug: Placebo — Placebo BID followed by assessment of safety, tolerability and efficacy on reducing the respiratory symptoms in patients.
  Arms: Placebo

SUMMARY:
This study evaluates the safety, tolerability and efficacy of Sarizotan in reducing respiratory abnormalities in Rett Syndrome in an initial double blind 24 week period followed by an open label treatment phase of up to 168 weeks (the latter for patients with no safety and tolerability issues).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, and efficacy of multiple doses of sarizotan in patients with Rett syndrome with respiratory abnormalities. The study participants will be randomized to either sarizotan between 2 and 10 mg bid or placebo bid, based on age and weight criteria.

All patients who have completed the final evaluations at Week 24 (Day 168) and have no safety or tolerability issues that would preclude continuing on the study medication and have been compliant with the trial requirements will have the option of continuing open-label treatment with Sarizotan for up to 168 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 10 kg
* Age ≥ 4 years
* Diagnosis of Rett syndrome based on consensus clinical criteria and patients with MECP2 duplications will not be eligible.
* Has at least 10 episodes of breathing dysrhythmia, defined by episodes ≥10 seconds of breath holding (apnea), per hour during cardiorespiratory monitoring
* Ability to take study medication provided either as capsules or combined with food/drink.
* Patient is cooperative, willing to complete all aspects of the study, and capable of doing so with assistance of a caregiver.

Exclusion Criteria:

* Meets any of the diagnostic exclusion criteria for Rett syndrome, Typical (Neul et al, 2010);
* Patient is participating in a clinical trial with another investigational drug
* Hypersensitivity to sarizotan or other 5-HT1a agonists;
* Current clinically significant (as determined by Investigator) cardiovascular, respiratory (e.g. severe asthma), gastrointestinal, renal, hepatic, hematologic or other medical disorders, in addition to those directly related to the patient's Rett syndrome;
* QTcF interval on the ECG is greater than 450 msec.
* Surgery planned during the study (except for insertion of gastrostomy tube);
* Severe diabetes mellitus or fatty acid oxidation disorder.
* Ophthalmologic history including any of the following conditions: albino patients, family history of hereditary retinal disease, retinitis pigmentosa, any active retinopathy or severe diabetic retinopathy.
* Females who are pregnant, breastfeeding, or of childbearing potential and not using a hormonal contraceptive.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Anand, MD, Study Director — Newron Pharmaceuticals
Locations (14):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, California
  - Rush University Medical Center, Chicago, Illinois
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Baylor College of Medicine, Houston, Texas
- South Metropolitan Health Service Fiona Stanley Hospital, Murdoch, Western Australia, Australia
- India (5):
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Vijaya Health Centre, Chennai, Tamil Nadu
  - P.D. Hinduja National Hospital and Medical Research Centre, Mumbai
  - Jaslok Hospital and Research centre, Mumbai
  - All India Institute of Medical Sciences, New Delhi
- Italy (2):
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena, Tuscany
  - U.O. Neuropsichiatria Infantile, Milan
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Background] Abdala AP, Dutschmann M, Bissonnette JM, Paton JF. Correction of respiratory disorders in a mouse model of Rett syndrome. Proc Natl Acad Sci U S A. 2010 Oct 19;107(42):18208-13. doi: 10.1073/pnas.1012104107. Epub 2010 Oct 4. PMID 20921395
- [Background] Abdala AP, Bissonnette JM, Newman-Tancredi A. Pinpointing brainstem mechanisms responsible for autonomic dysfunction in Rett syndrome: therapeutic perspectives for 5-HT1A agonists. Front Physiol. 2014 May 30;5:205. doi: 10.3389/fphys.2014.00205. eCollection 2014. PMID 24910619
- [Background] Abdala AP, Lioy DT, Garg SK, Knopp SJ, Paton JF, Bissonnette JM. Effect of Sarizotan, a 5-HT1a and D2-like receptor agonist, on respiration in three mouse models of Rett syndrome. Am J Respir Cell Mol Biol. 2014 Jun;50(6):1031-9. doi: 10.1165/rcmb.2013-0372OC. PMID 24351104
- [Background] Adams JA, Zabaleta IA, Stroh D, Sackner MA. Measurement of breath amplitudes: comparison of three noninvasive respiratory monitors to integrated pneumotachograph. Pediatr Pulmonol. 1993 Oct;16(4):254-8. doi: 10.1002/ppul.1950160408. PMID 8265274
- [Background] Bloch KE, Li Y, Sackner MA, Russi EW. Breathing pattern during sleep disruptive snoring. Eur Respir J. 1997 Mar;10(3):576-86. PMID 9072988
- [Background] Brouillette RT, Morrow AS, Weese-Mayer DE, Hunt CE. Comparison of respiratory inductive plethysmography and thoracic impedance for apnea monitoring. J Pediatr. 1987 Sep;111(3):377-83. doi: 10.1016/s0022-3476(87)80457-2. PMID 3625404
- [Background] Byard RW. Forensic issues and possible mechanisms of sudden death in Rett syndrome. J Clin Forensic Med. 2006 Feb;13(2):96-9. doi: 10.1016/j.jcfm.2005.08.013. Epub 2005 Nov 2. PMID 16263320
- [Background] Cantineau JP, Escourrou P, Sartene R, Gaultier C, Goldman M. Accuracy of respiratory inductive plethysmography during wakefulness and sleep in patients with obstructive sleep apnea. Chest. 1992 Oct;102(4):1145-51. doi: 10.1378/chest.102.4.1145. PMID 1395758
- [Background] Clarenbach CF, Senn O, Brack T, Kohler M, Bloch KE. Monitoring of ventilation during exercise by a portable respiratory inductive plethysmograph. Chest. 2005 Sep;128(3):1282-90. doi: 10.1378/chest.128.3.1282. PMID 16162719
- [Background] Collop NA, Anderson WM, Boehlecke B, Claman D, Goldberg R, Gottlieb DJ, Hudgel D, Sateia M, Schwab R; Portable Monitoring Task Force of the American Academy of Sleep Medicine. Clinical guidelines for the use of unattended portable monitors in the diagnosis of obstructive sleep apnea in adult patients. Portable Monitoring Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2007 Dec 15;3(7):737-47. PMID 18198809
- [Background] Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0, May 28, 2009 (v4.03 June 14, 2010), U.S. Department of Health and Human Services.
- [Background] FitzGerald PM, Jankovic J, Percy AK. Rett syndrome and associated movement disorders. Mov Disord. 1990;5(3):195-202. doi: 10.1002/mds.870050303. PMID 2388636
- [Background] Guy W (Ed). Clinical Global Impressions. In ECDEU Assessment Manual for Psychopharmacology, revised, U.S. Department of Health, Education and Welfare Pub. No. (ADM) 76-338. Rockville, MD: NIMH, 1976, 217-222.
- [Background] Hammer J, Newth CJ, Deakers TW. Validation of the phase angle technique as an objective measure of upper airway obstruction. Pediatr Pulmonol. 1995 Mar;19(3):167-73. doi: 10.1002/ppul.1950190305. PMID 7792119
- [Background] Julu PO, Kerr AM, Hansen S, Apartopoulos F, Jamal GA. Immaturity of medullary cardiorespiratory neurones leading to inappropriate autonomic reactions as a likely cause of sudden death in Rett's syndrome. Arch Dis Child. 1997 Nov;77(5):464-5. doi: 10.1136/adc.77.5.463c. No abstract available. PMID 9487980
- [Background] Julu PO, Kerr AM, Apartopoulos F, Al-Rawas S, Engerstrom IW, Engerstrom L, Jamal GA, Hansen S. Characterisation of breathing and associated central autonomic dysfunction in the Rett disorder. Arch Dis Child. 2001 Jul;85(1):29-37. doi: 10.1136/adc.85.1.29. PMID 11420195
- [Background] Julu PO, Engerstrom IW, Hansen S, Apartopoulos F, Engerstrom B, Pini G, Delamont RS, Smeets EE. Cardiorespiratory challenges in Rett's syndrome. Lancet. 2008 Jun 14;371(9629):1981-3. doi: 10.1016/S0140-6736(08)60849-1. No abstract available. PMID 18555901
- [Background] Katz DM, Dutschmann M, Ramirez JM, Hilaire G. Breathing disorders in Rett syndrome: progressive neurochemical dysfunction in the respiratory network after birth. Respir Physiol Neurobiol. 2009 Aug 31;168(1-2):101-8. doi: 10.1016/j.resp.2009.04.017. Epub 2009 Apr 24. PMID 19394452
- [Background] Kerr AM, Armstrong DD, Prescott RJ, Doyle D, Kearney DL. Rett syndrome: analysis of deaths in the British survey. Eur Child Adolesc Psychiatry. 1997;6 Suppl 1:71-4. PMID 9452925
- [Background] Khwaja OS, Ho E, Barnes KV, O'Leary HM, Pereira LM, Finkelstein Y, Nelson CA 3rd, Vogel-Farley V, DeGregorio G, Holm IA, Khatwa U, Kapur K, Alexander ME, Finnegan DM, Cantwell NG, Walco AC, Rappaport L, Gregas M, Fichorova RN, Shannon MW, Sur M, Kaufmann WE. Safety, pharmacokinetics, and preliminary assessment of efficacy of mecasermin (recombinant human IGF-1) for the treatment of Rett syndrome. Proc Natl Acad Sci U S A. 2014 Mar 25;111(12):4596-601. doi: 10.1073/pnas.1311141111. Epub 2014 Mar 12. PMID 24623853
- [Background] Konno K, Mead J. Measurement of the separate volume changes of rib cage and abdomen during breathing. J Appl Physiol. 1967 Mar;22(3):407-22. doi: 10.1152/jappl.1967.22.3.407. No abstract available. PMID 4225383
- [Background] Landon C. Respiratory monitoring: Advantages of inductive plethysmography over impedance pneumograpy. VivoMetrics, VMLA-039-02, 2003.
- [Background] Leino K, Nunes S, Valta P, Takala J. Validation of a new respiratory inductive plethysmograph. Acta Anaesthesiol Scand. 2001 Jan;45(1):104-11. doi: 10.1034/j.1399-6576.2001.450116.x. PMID 11152021
- [Background] Loube DI, Andrada T, Howard RS. Accuracy of respiratory inductive plethysmography for the diagnosis of upper airway resistance syndrome. Chest. 1999 May;115(5):1333-7. doi: 10.1378/chest.115.5.1333. PMID 10334149
- [Background] Neul JL, Fang P, Barrish J, Lane J, Caeg EB, Smith EO, Zoghbi H, Percy A, Glaze DG. Specific mutations in methyl-CpG-binding protein 2 confer different severity in Rett syndrome. Neurology. 2008 Apr 15;70(16):1313-21. doi: 10.1212/01.wnl.0000291011.54508.aa. Epub 2008 Mar 12. PMID 18337588
- [Background] Neul JL, Kaufmann WE, Glaze DG, Christodoulou J, Clarke AJ, Bahi-Buisson N, Leonard H, Bailey ME, Schanen NC, Zappella M, Renieri A, Huppke P, Percy AK; RettSearch Consortium. Rett syndrome: revised diagnostic criteria and nomenclature. Ann Neurol. 2010 Dec;68(6):944-50. doi: 10.1002/ana.22124. PMID 21154482
- [Background] Neul JL, Glaze DG, Percy AK, Feyma T, Beisang A, Dinh T, Suter B, Anagnostou E, Snape M, Horrigan J, Jones NE. Improving Treatment Trial Outcomes for Rett Syndrome: The Development of Rett-specific Anchors for the Clinical Global Impression Scale. J Child Neurol. 2015 Nov;30(13):1743-8. doi: 10.1177/0883073815579707. Epub 2015 Apr 20. PMID 25895911
- [Background] Sackner MA, Watson H, Belsito AS, Feinerman D, Suarez M, Gonzalez G, Bizousky F, Krieger B. Calibration of respiratory inductive plethysmograph during natural breathing. J Appl Physiol (1985). 1989 Jan;66(1):410-20. doi: 10.1152/jappl.1989.66.1.410. PMID 2917945
- [Background] Weng SM, Bailey ME, Cobb SR. Rett syndrome: from bed to bench. Pediatr Neonatol. 2011 Dec;52(6):309-16. doi: 10.1016/j.pedneo.2011.08.002. Epub 2011 Nov 6. PMID 22192257
- [Derived] Gualniera L, Singh J, Fiori F, Santosh P. Emotional Behavioural and Autonomic Dysregulation (EBAD) in Rett Syndrome - EDA and HRV monitoring using wearable sensor technology. J Psychiatr Res. 2021 Jun;138:186-193. doi: 10.1016/j.jpsychires.2021.03.052. Epub 2021 Apr 7. PMID 33862302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 sites in 5 countries. Enrollment occurred from 26-Oct-2016 through February 2019 . An analysis was planned when the primary efficacy data at Week 24 were available for all patients (06 August 2019 - last patient last visit for double-blind part of the study). Patients without safety and tolerability issues continued in the open label with sarizotan for an additional 24 weeks and then another 48 weeks if no safety issues were present.
Pre-assignment Details: A total of 198 patients were screened, of which 69 (34.8%) patients were screen failures.
  A total of 129 patients were randomized in the study. A total of 128 patients were exposed to at least one dose of IMP, with placebo ITT group (40) vs safety pop (39).
Groups:
- Placebo: Placebo bid for 24 wks DB
Period: Overall Study
Arm/Group | Sarizotan Low Dose | Sarizotan High Dose | Placebo
Started | 33 | 56 | 40
Completed | 27 | 46 | 36
Not Completed | 6 | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo BID
- Total: Total of all reporting groups
Arm/Group | Sarizotan Low Dose | Sarizotan High Dose | Placebo | Total
Number analyzed (Participants) | 33 | 56 | 40 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 35 | 27 | 85
  Between 18 and 65 years | 10 | 21 | 13 | 44
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.23 (7.195) | 15.55 (9.362) | 14.13 (9.155) | 14.51 (8.780)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 56 | 40 | 129
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 4 | 13
  Not Hispanic or Latino | 29 | 51 | 36 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 16 | 13 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 1 | 3 | 5
  White | 23 | 37 | 22 | 82
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 19 | 11 | 41
  Italy | 8 | 13 | 9 | 30
  United Kingdom | 5 | 10 | 6 | 21
  Australia | 1 | 0 | 2 | 3
  India | 8 | 14 | 12 | 34
Duration of Rett syndrome [Mean (Standard Deviation); unit: months] | 87.90 (72.536) | 97.18 (72.922) | 73.94 (65.800) | 87.94 (70.696)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Respiratory Abnormality in Patients With Rett Syndrome
Description: Measured as the percent change in the number of apnea episodes per hour during awake time, calculated using an ambulatory data acquisition system (BioRadioTM) as part of home monitoring procedure. BioRadioTM record specific respiratory and cardiac parameters.
Time Frame: Baseline up to week 24
Population: The ITT population included all patients who were randomized to treatment. This population was used for all efficacy analysis.
Measure: Least Squares Mean (Standard Error); unit: % of change in mean counts per hr
Arm/Group | Sarizotan Low Dose | Sarizotan High Dose | Placebo
Number analyzed (Participants) | 33 | 56 | 40
% of change in mean counts per hr | 1.54 (10.1228) | 13.211 (7.5075) | 18.503 (8.441)
Statistical Analysis 1: Comparison: Sarizotan High Dose vs Placebo; Primary inferential comparison between treatment groups used a restricted maximum likelihood (REML)-based, mixed-effects repeated measures model approach (MMRM) with 95% CI for the difference between treatment groups for % change from baseline in the number of apnea episodes. Model included % change from baseline as response, the fixed, categorical effects of treatment group, visit, treatment group-by-visit interaction, and the continuous terms age and baseline value as covariate; Test type: Superiority; p = 0.6411, Mixed Models Analysis; Mean Difference (Final Values) = -5.292, 95% CI 2-sided [-27.741 to 17.157], Standard Error of Mean 11.3184
Statistical Analysis 2: Comparison: Sarizotan Low Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2011, Mixed Models Analysis; Mean Difference (Final Values) = -16.966, 95% CI 2-sided [-43.119 to 9.186], Standard Error of Mean 13.1869

2. Secondary Outcome: Efficacy of Sarizotan Assessed by the Caregiver-rated Impression of Change
Description: Caregiver-rated Impression of Change (CIC): 7-point scale requiring the caregiver to rate how much the patient's illness has improved or worsened relative to the baseline state.
  7-point Likert-type scale for which ratings range from 1 = very much improved to 7 = very much worse, with 4 = no change. This caregiver-rated measure considered activities, behavior, mood and functioning. This rating was performed in consultation with the study Investigator but was based largely on the caregivers' evaluation during the reporting period. The single rating of the CIC was to be based on changes in the following domains: • Activities (watching TV, interest in conversations around her, cooperation during toileting, dressing/bathing, etc.), • Communication (verbal or by eye movements, hand movements, or head movements), • Behavior (agitation, refusal to feed, scratching, social avoidance), • Participation in family/outdoor/social events)
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sarizotan Low Dose | Sarizotan High Dose | Placebo
Number analyzed (Participants) | 33 | 56 | 40
score on a scale | 3.6 (0.67) | 3.5 (1.12) | 3.4 (0.79)

ADVERSE EVENTS:
Time Frame: AEs will be collected, from the time of signing of Informed Consent to the end of the safety follow-up period (14 days after last dose of study medication at 24 weeks). In addition, all subjects will be followed up for 30 days after last dose for SAEs, up to a total of 28 weeks.
Description: Analysis population = safety population defined as all patients randomized and exposed to at least one dose of IMP. One patient randomized to placebo treatment did not receive IMP, hence placebo ITT group (40) vs safety pop (39).
  Classification of the Event: Classify the event as either serious or non-serious Description of Signs or Symptoms: Whenever possible, record a specific diagnosis for the event Start/stop date Intensity (mild, moderate, severe) Causality Action taken with IMP
Groups:
- Sarizotan Low Dose: 2 mg or 5 mg bid based on age and weight criteria for 24 wks DB
  2 mg bid (4 to <13 years; ≥13 years of age and weighing <25 kg
  5 mg bid (≥13 years of age and weighing ≥25 kg)
  Assessment of safety, tolerability and efficacy on reducing the respiratory symptoms in patients.
- Sarizotan High Dose: 5 mg or 10 mg bid based on age and weight criteria for 24 wks DB
  5 mg bid (4 to <13 years; ≥13 years of age and weighing <25 kg
  10 mg bid (≥13 years of age and weighing ≥25 kg)
  Assessment of safety, tolerability and efficacy on reducing the respiratory symptoms in patients.
- Placebo: Placebo bid respectively
  Placebo: placebo BID followed by assessment of safety, tolerability and efficacy on reducing the respiratory symptoms in patients.
Arm/Group | Sarizotan Low Dose | Sarizotan High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/56 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/33 | 10/56 | 5/39
Other Adverse Events (participants affected / at risk) | 25/33 | 46/56 | 30/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarizotan Low Dose (N=33) | Sarizotan High Dose (N=56) | Placebo (N=39)
Seizure (Nervous system disorders) | 1 (1) | 0 | 0
Gingival Hypertrophy (Gastrointestinal disorders) | 1 (1) | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0
Gingivitis (Infections and infestations) | 1 (1) | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0
Acute respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Somnolence (Nervous system disorders) | 0 | 2 (2) | 1 (1)
Change in seizure presentation (Nervous system disorders) | 0 | 1 (1) | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 0 | 1 (1) | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1 (1) | 0
Pneumonia (Infections and infestations) | 0 | 1 (1) | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarizotan Low Dose (N=33) | Sarizotan High Dose (N=56) | Placebo (N=39)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4)
Seizure (Nervous system disorders) | 8 (8) | 15 (15) | 5 (5)
Somnolence (Nervous system disorders) | 2 (2) | 10 (10) | 6 (6)
Psychomotor hyperactivity (Nervous system disorders) | 4 (4) | 1 (1) | 3 (3)
Dystonia (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 0
Sleep Disorder (Psychiatric disorders) | 3 (3) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
No efficacy evaluation was performed for the open label extension, as the study was terminated prematurely by the Sponsor based on lack of demonstrated efficacy in the double-blind period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT02790034/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT02790034/SAP_001.pdf